CLINICAL TRIAL: NCT05379400
Title: Cardiometabolic Biomarker Improvements Associated With Reduction in Air Pollution Exposure Via Home Air Filtration
Brief Title: Cleaner Air for Better Cardiac Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-00045
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portable Air Cleaner (PAC) group (Experimental): This study will utilize a portable air cleaner as an intervention for the potential reduction of air pollution-associated inflammation. This commercially available device has no significant risks. The researchers plan to use a commercially available PAC with a "true HEPA" filter for the true arm.
  Interventions: Other: Portable air cleaner (PAC)
- Sham Portable Air Cleaner (PAC) group (Sham Comparator): For the sham arm, the same model will be used with HEPA filter removed, and has identical appearance and sound. The researchers will use a PAC designed to filter air in rooms up to approximately 350 ft2, with minimal noise on the lowest setting.
  Interventions: Other: Sham Portable air cleaner (PAC)

INTERVENTIONS:
Other: Portable air cleaner (PAC) — Commercially available Portable air cleaners (PAC) contain carbon filters that reduce volatile organic carbons and can reduce odors. Because of this, the researchers will remove the carbon filters from all air purifiers to preserve blinding. This will be done by unblinded research staff and devices will be labelled with an ID number to preserve blinding of the rest of the research team.
  Arms: Portable Air Cleaner (PAC) group
Other: Sham Portable air cleaner (PAC) — Sham Portable air cleaner (PAC) are commercially available portable air cleaners with the carbon filters and the HEPA filters removed. This will be done by unblinded research staff and devices will be labelled with an ID number to preserve blinding of the rest of the research team.
  Arms: Sham Portable Air Cleaner (PAC) group

SUMMARY:
This pilot project is a randomized, double-blind, sham-controlled trial investigating whether in-home air pollution reductions using portable air cleaners (PACs) can decrease circulating concentrations of biomarkers of inflammation. Using both a targeted approach to study the established biomarker TNFa and an exploratory approach with a commercially available proteomic panel, the researchers will measure concentrations of biomarkers before and after four weeks of home PAC use in a cohort of 74 adults with hypertension recruited from NYU outpatient clinical settings. Participants will also track home blood pressure measurements for additional exploratory analysis of potential mediation of PAC-associated decreases in blood pressure by biomarker concentration changes.

DETAILED DESCRIPTION:
In Aim 1, the researchers will evaluate associations with PAC use with a priori specified biomarker of inflammation, tumor necrosis factor alpha (TNFα). The researchers will determine if 4 weeks of home air filtration with PACs compared to sham is associated with significant reductions in TNFα concentrations when measured before and after intervention. Blood samples will be collected from 74 study participants before and after 4 weeks of PAC use (true and sham) for biomarker concentration measurement. In Aim 2, the researchers will determine if reductions in fine particulate matter (<2.5 μm in diameter, PM2.5) as a continuous variable are associated with significant reductions TNFα concentrations over a four-week period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥18 years old
* Participant and members of household are reported to be non-smokers (defined as no household members are currently known to smoke cigarettes or use other tobacco products including e-cigarettes)
* Participant is to understand/speak English or Spanish
* Participant can understand study procedures and give informed consent
* Participant has stable hypertension: no medication changes in prior 30 days, systolic BP <160 mm Hg and either ≥ 130 mm Hg without antihypertensive medications, or diagnosis of hypertension in medical records
* Able to measure home blood pressure twice daily
* Able to participate in video conference for home equipment setup
* Able to visit clinic for blood draws before and after the study period
* Do not intend to sleep anywhere outside of primary bedroom for more than 48 consecutive hours or a total of 7 days during the study period.
* Ability to lift, or access to assistance with lifting, 20 lb to set up PAC in bedroom.

Exclusion Criteria:

* Participants who are unable to provide a minimum of at least one blood pressure measurement per day
* Participants with average home blood pressure monitor readings of a systolic blood pressure (SBP) >160 mmHg over any 10-day period during the study. This will be considered evidence of uncontrolled hypertension and will require study termination.
* Participants with known coronary artery disease
* Participants with known systemic inflammatory conditions (such as rheumatoid arthritis, inflammatory bowel disease, cancer)
* Participants currently taking any anti-inflammatory medications or medications that target inflammatory cytokines
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Newman, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Jonathan.Newman@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 participants were enrolled, n=2 did not start the study.
Period: Overall Study
Arm/Group | Portable Air Cleaner (PAC) Group | Sham Portable Air Cleaner (PAC) Group
Started | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portable Air Cleaner (PAC) Group | Sham Portable Air Cleaner (PAC) Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.8) | 57.8 (11) | 58.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 12 | 8 | 20
  Unknown or Not Reported | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 8 | 10 | 18
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Circulating Concentration of Tumor Necrosis Factor Alpha (TNFα)
Description: Circulating concentrations of TNFα will be measured using the Olink Explore 384 Cardiometabolic panel for this a priori specified analysis.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Portable Air Cleaner (PAC) Group | Sham Portable Air Cleaner (PAC) Group
Number analyzed (Participants) | 22 | 22
percent change | -1.03 (8.35) | 2 (3.69)

2. Secondary Outcome: Change in Indoor Particulate Matter < 2.5 um in Diameter (PM2.5) Concentration
Description: Commercially available Particulate Matter (PM) monitors will record indoor PM2.5 concentrations using dual (backup) sensors, which store measurements on internal SD cards
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: micrograms per cubic meter air (μ/m3)
Arm/Group | Portable Air Cleaner (PAC) Group | Sham Portable Air Cleaner (PAC) Group
Number analyzed (Participants) | 22 | 22
micrograms per cubic meter air (μ/m3) | 2.698 (2.483) | 11.751 (20.93)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: Self-report.
Arm/Group | Portable Air Cleaner (PAC) Group | Sham Portable Air Cleaner (PAC) Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT05379400/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT05379400/ICF_000.pdf